CLINICAL TRIAL: NCT06086886
Title: A Phase 1, Double-blinded, Randomized, Placebo-controlled, First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Doses of BMS-986454 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability and Drug Levels of BMS-986454 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM055-1001; U1111-1270-3670 (Registry Identifier: WHO)
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Healthy Participants
Keywords: Pharmacokinetics; Pharmacodynamics; Healthy Participants; BMS-986454; First-in-human; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BMS-986454 (Experimental)
  Interventions: Drug: BMS-986454
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986454 — Specified dose on specified days
  Arms: BMS-986454
Other: Placebo — Specified dose on specified days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of BMS-986454 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are healthy as determined by the investigator based on review of medical history, physical examinations, 12-lead ECGs, and clinical laboratory tests obtained during the screening period.
* Participant is willing and able to adhere to the study visit schedule and other protocol requirements.
* A negative test for COVID-19, which will be performed in the manner mandated by the clinical site where this study is being conducted, at screening and admission.

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, 12-lead ECG, or clinical laboratory tests beyond what is consistent with a healthy population in the region in which the study is conducted.
* Participant was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or 5 half-lives of that investigational drug, if known (whichever is longer).
* Inability to be venipunctured or tolerate venous access.

Note: Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to approximately 4 months
Number of participants with severe adverse events (SAEs) | Up to approximately 4 months
Number of participants with physical examination abnormalities | Up to approximately 4 months
Number of participants with vital sign abnormalities | Up to approximately 4 months
Number of participants with electrocardiogram (ECG) abnormalities | Up to approximately 4 months
Number of participants with clinical laboratory abnormalities | Up to approximately 4 months

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) | Up to approximately 3 months
Time of maximum observed serum concentration (Tmax) | Up to approximately 3 months
Area under concentration time curve from time 0 to time of last quantifiable concentration [AUC(0-T)] | Up to approximately 3 months
Incidence of anti-drug antibody (ADA) formation | Up to approximately 3 months
Absolute Bioavailability (F) of BMS-986454 | Up to approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United Kingdom (2):
  - Local Institution - 0002, London, Greater London
  - Local Institution - 0001, Nottingham

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com